CLINICAL TRIAL: NCT05474326
Title: Amniotic Fluid Index and Fetal Doppler Indices Measurment After Application of Intermittent Pneumatic Compression Device on Lower Limbs in Pregnant Women With Oligohydramnios
Brief Title: Effect of Intermittent Pneumatic Compression Device of Lower Limbs in Oligohydramnios
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Inshirah Sgayer, Dr. Inshirah Sgayer, Western Galilee Hospital-Nahariya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9999
Record Dates: First submitted 2021-12-07; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Oligohydramnios; Amniotic Fluid; Disorder
MeSH Terms: conditions — Oligohydramnios

STUDY DESIGN:
Intervention Model Description: The Kendall SCD™ 700 Smart Compression™ Controller is an intermittent pneumatic compression (IPC) device application of this intermittent pneumatic pressure device on lower limbs in women with oligohydramnios and its effect on maternal uterine artery doppler, fetal umbilical artery doppler, middle cerebral artery doppler
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- pregnant women with idiopathic oligohydramnios (Experimental): women with singleton pregnancy between 32-41 weeks oligohydramnios diagnosed by ultrasound by the amniotic fluid index (AFI) method oligohydramnios is diagnosed if AFI index is less than 5 cm
  Interventions: Device: intermittent pneumatic pressure device (Kendall SCD™ 700 Smart Compression™ System)

INTERVENTIONS:
Device: intermittent pneumatic pressure device (Kendall SCD™ 700 Smart Compression™ System) — application of intermittent pneumatic pressure device (Kendall SCD™ 700 Smart Compression™ System) on lower limbs and its effect on fetal and maternal doppler and amniotic fluid index in women with oligohydramnios. the compression system will be applicated on lower limbs for one hour in which it will produce intermittent compression on lower limbs. amniotic fluid amnout assessment will be done after this including doppler studies in order to detect any change in amniotic fluid amount or dopper.

SUMMARY:
the study will examine the effect of application of intermittent pneumatic pressure device on lower limbs on the amniotic fluid amount and fetal doppler indices in women with oligohydramnios

DETAILED DESCRIPTION:
oligohydramnios is diagnosed based on ultrasonographic finding of amniotic fluid index less than 5 cm.

Etiologies of oligohydramnios includes infection with viruses such as rubella, cytomegalo virus or parasites such as toxoplasma. other etiologies includes rupture of membranes or fetal malformatios especially urinary tract anomalies. in addition, placental insuffiency may lead to oligohydramnios and can be diagnosed through abnormal doppler measures in the umbilical and middle cereberal arteries. when these etiologies are excluded oligohydramnios is considered to be idiopathic.

The Kendall SCD™ 700 Smart Compression™ Controller is an intermittent pneumatic compression (IPC) device which delivers compression to the legs and feet to aid in the prevention of Venous Thromboembolism in at-risk patient.

previous studies had shown that intermittent pneumatic compression device may increase cardiac output through preload increase.

the study hypothesis that after the application of IPC there will be an improvement in the preload and cardiac which will lead to an increase in placental perfusion and eventually will lead to increase in amniotic fluid amount and improvement in fetal doppler measurement.

the study will include women with a diagnosis of idiopathic oligohydramnios between 32-41 weeks and who will agree to participate in the study the diagnosis of idiopathic oligohydramnios is based on ultrasonographic diagnosis of amniotic fluid index of less than 5 cm after exclusion of other etiologies.

The amniotic fluid index (AFI) is measured by dividing the uterus into four imaginary quadrants. The linea nigra is used to divide the uterus into right and left halves.The umbilicus serves as the dividing point for the upper and lower halves.

The transducer is kept parallel to the patient's longitudinal axis and perpendicular to the floor. The deepest, unobstructed, vertical pocket of fluid is measured in each quadrant in centimeters. The four pocket measurements are then added to calculate the AFI. Normal AFI values range from 5 to 25 cm. women with AFI<5 cm will be diagnosed with oligohydramnios.

The amniotic fluid fluid index (AFI) will be measured in centemeters before the application of IPC the IPC device will be applied to the lower limbs for one hour after this a repeated measurement of AFI in centemeters will be performed.

additionally, doppler studies will be performed. Pulsed wave high-resolution color doppler uhrasonography will be used to identify and to obtain blood flow velocity waveforms from the following vessels: (1) umbilical artery, from a free loop of theumbilical cord; (2) middle cerebral artery, from the main vessel identified branching from the circle of Willis at the anterior wing of the sphenoid; (3) renal artery, from the vessel identified branching from the abdominal aorta into the hilum of the kidney, and (4) maternal uterine artery, from the vessel branching from the internal iliac artery on the placental side.

In all vessels the pulsatility index will be calculated with the mean of at least three consecutive waveforms used for analysis.

ELIGIBILITY:
Inclusion Criteria:

pregnant women with a diagnosis of oligohydramnios

Exclusion Criteria:

* fetal malformation
* rupture of membranes
* documented viral infection with rubella, cytomegalovirus, herpes simplex, toxoplsma in pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 30 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
pulsatility index in maternal uterine artery | one hour
  Pulsed wave high-resolution color Doppler uhrasonography will be used to identify and to obtain blood flow velocity waveforms. PI will be calculated from the difference in the systolic and diastolic flow velocity divided by the mean flow velocity baseline PI of the maternal uterine artery will be calculated before the application of IPC on lower maternal limbs PI of the maternal uterine artery will be re-calculated after the application of IPC on lower maternal limbs for one hour
pulsatility index in fetal umbilical artery | one hour
  Pulsed wave high-resolution color Doppler uhrasonography will be used to identify and to obtain blood flow velocity waveforms. PI will be calculated from the difference in the systolic and diastolic flow velocity divided by the mean flow velocity baseline PI of the fetal umbilical artery will be calculated before the application of IPC on lower maternal limbs PI of the fetal umbilical artery will be re-calculated after the application of IPC on lower maternal limbs for one hour
pulsatility index in fetal middle cerebral artery | one hour
  Pulsed wave high-resolution color Doppler uhrasonography will be used to identify and to obtain blood flow velocity waveforms. PI will be calculated from the difference in the systolic and diastolic flow velocity divided by the mean flow velocity baseline PI of the fetal middle cerebral artery will be calculated before the application of IPC on lower maternal limbs PI of the fetal middle cerebral artery will be re-calculated after the application of IPC on lower maternal limbs for one hour
pulsatility index in fetal renal artery | one hour
  Pulsed wave high-resolution color Doppler uhrasonography will be used to identify and to obtain blood flow velocity waveforms. PI will be calculated from the difference in the systolic and diastolic flow velocity divided by the mean flow velocity baseline PI of the fetal renal artery will be calculated before the application of IPC on lower maternal limbs PI of the fetal renal artery will be re-calculated after the application of IPC on lower maternal limbs for one hour
amniotic fluid index | one hour
  basline amniotic fluid index (AFI in centemeters) will be calculated before the application of IPC on lower maternal limbs amniotic fluid index (AFI in centemeters) will be re-calculated after the application of IPC on lower maternal limbs for one hour

CONTACTS AND LOCATIONS:
Overall Officials: inshirah sgayer, MD, Principal Investigator — GALILEE MEDICAL CENTER ISRAEL